CLINICAL TRIAL: NCT06093347
Title: Feasibility Study to Evaluate a New Wearable Wireless Device for Monitoring Central Apnoeas in Infants and Children
Brief Title: Central Apnoea Monitor Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Collaborators: Sheffield Hallam University (Other)
Responsible Party: Sponsor
Other Study IDs: SCH-2708
Record Dates: First submitted 2023-09-25; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-09

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An initial small study on 15 children that are already being investigated for central sleep apnoea in the sleep unit at Sheffield Children's Hospital. The central apnoea monitor will be placed around the child's abdomen overnight alongside the sensors already being used for the clinical sleep study and the signals from the two systems will be compared to evaluate the accuracy of the new device.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been referred for a cardio-respiratory polygraphy sleep study.
* Patients aged 1 month up to 5 years old.

Exclusion Criteria:

* Subjects whose parents/legal guardians/carers are not fluent in English, or who have special communication needs.
* Child anticipated to become distressed with additional sensor.
* Child too clinically unwell to take part (as decided by clinical staff).

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children admitted to the Sleep Unit at Sheffield Children's Hospital with suspected sleep apnoea
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
The accuracy of the system in 15 patients, when compared with the gold standard measurement system | 24 hours
The acceptability of the sensor to the child as viewed by the parent (and child) | End of study
  As measured by researcher designed questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Facility, Sheffield Children's Hospital, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No